CLINICAL TRIAL: NCT04812184
Title: Adhesive Tape Placement on Patients' Masks in the Emergency Department Increases Compliance of Proper Face Mask Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Nicholas Pettit, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUMASKstudy
Record Dates: First submitted 2021-03-17; First posted 2021-03-23 (Actual); Results first posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Surgical Tape to bridge of nose (Experimental): placed a piece of tape to the bridge of the nose, adhering a face mask to the patient's face
  Interventions: Device: Tape Face Mask
- Standard of care (No Intervention): Patients given a mask with no intervention to the mask

INTERVENTIONS:
Device: Tape Face Mask — Adding tape to face mask
  Arms: Surgical Tape to bridge of nose

SUMMARY:
Methods 123 patients were enrolled in a randomized controlled trial at Eskenazi Hospital from April 2020 until October 2020. We permitted patients to either use their own mask (due to low resources institutionally) or we provided a surgical/cloth mask (early on relied on donated cloth masks for patients). Patients were randomized to a control (no tape over the mask/nose) or to the intervention (placing tape over the bridge of the nose of the face mask). Patients were evaluated at 30- and 60- minute intervals to assess for proper mask usage.

DETAILED DESCRIPTION:
Study Design and Setting:

This study is a randomized control trial at Eskenazi Hospital ED from April 2020 until October 2020. Eskenazi Hospital is a busy, urban, academic hospital, level 1 trauma center, in downtown Indianapolis. Here we serve a racially diverse, underserved population, with over 100,000 annual ED visits. This work was approved by the Indiana University Institutional Review Board (protocol #2004425945).

Selection of Participants:

All patients presenting to the ED were screened for enrollment in this study by trained research personnel. All patients are required to wear facial coverings while in the ED, and after screening patients based on the exclusion criteria provided below, patients were offered enrollment in the study. Patients were randomly identified by their bed location in the ED via a random number generator. Patients were excluded from the study for: (1) pregnant; (2) prisoner; (3) not English or Spanish speaking (currently a large cohort of ethnic Latino/Latina/Hispanic are utilizing the ED and we can use interpreters to interpret for enrollment); (4) intoxicated or decompensated psychiatric illness; (5) presenting to the ED with a life-threatening condition; (6) allergic to standard tape and/or tegaderm. Patient consent was obtained if an individual agreed to participate in the study.

Interventions:

All patients included in this study were approached and offered enrollment in a study for addressing PPE. The control arm consisted of no active intervention, with the treatment arm placing standard surgical tape over the bridge of the nose to adhere the top of the mask to the bridge of the nose, thereby creating a physical barrier from removing the mask from the face. Patients were reevaluated at 30 minutes and 60 minutes after enrollment to assess for proper mask compliance.

Measurements: Assuming 50% current compliance, 58 patients per arm were needed to have an 80% power to detect a 25% difference assuming a two-sided chi-square test and alpha = 0.05.

Outcomes:

The primary outcome of this trial is proper mask utilization upon reevaluation at 30 and 60 minutes, with the mask at/under the chin, meanwhile completely covering the mouth and nose). Secondary outcomes of this trial were comparing the primary demographic and visit related covariates on initial screening, including age, sex, race/ethnicity, past medical history, social history, chief complaint, and disposition (admission vs. discharge).

Analysis:

Patient demographics and characteristics were compared between the control and treatment groups. To test for differences between groups, Microsoft excel statistical package was utilized, and the Chi-square test was used for categorical variables and the Wilcoxon test for continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* presenting to the emergency department during the covid-19 pandemic
* older than 18 years of age

Exclusion Criteria:

* pregnant
* prisoner
* not english speaking
* not intoxicated or decompensated psychiatric illness
* not critically ill
* not allergic to standard tape and/or tegaderm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Pettit, Principal Investigator — Indiana University
Locations (1):
- Eskenazi Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
data available upon request

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting to the ED were screened for enrollment by trained research personnel when one of the study authors was working. This study was an open-label randomized control trial at Eskenazi Hospital ED from April 2020 to October 2020.
Period: Overall Study
Arm/Group | Surgical Tape to Bridge of Nose | Standard of Care
Started | 60 | 63
Completed | 60 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: Patients given a mask with no intervention to the mask, unless they had their own mask
- Total: Total of all reporting groups
Arm/Group | Surgical Tape to Bridge of Nose | Standard of Care | Total
Number analyzed (Participants) | 60 | 63 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 5 | 62
  >=65 years | 3 | 58 | 61
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41 [30.5 to 55.3] | 42 [31.5 to 55] | 41 [31 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 36 | 61
  Male | 35 | 27 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 35 | 67
  White | 26 | 24 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 60 | 63 | 123
mask type [Count of Participants; unit: Participants]
  Home mask | 35 | 46 | 81
  Provided mask | 25 | 17 | 42

OUTCOME MEASURES:

1. Primary Outcome: Proper Face Mask Use up to 60 Minutes
Description: The primary outcome of this trial is proper mask utilization upon reevaluation up to 60 minutes (with the mask at/under the chin, meanwhile completely covering the mouth and nose). At these time point a trained observer enters the room and observes the patient's face covering and its location on the face (correct, chin exposed, nose exposed, not on at all).
Time Frame: 60 minutes on Day 1
Population: Overall number of participants analyzed less than total 123. 2 patients were discharged prior to the 60 minute reevaluation from the standard of care group.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Tape to Bridge of Nose | Standard of Care
Number analyzed (Participants) | 58 | 61
Participants | 58 | 52

ADVERSE EVENTS:
Time Frame: within the single emergency department visit
Arm/Group | Surgical Tape to Bridge of Nose | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/63
Other Adverse Events (participants affected / at risk) | 0/60 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT04812184/Prot_SAP_000.pdf